CLINICAL TRIAL: NCT06837857
Title: Imaging, Cognition, and Opioids in Older Adults With Chronic Pain (I-COAP) Trial
Brief Title: Prescription Opioids, Brain Structure, and Cognition in Older Adults With Chronic Pain
Acronym: I-COAP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Nafisseh S. Warner, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 24-008096
Record Dates: First submitted 2025-02-06; First posted 2025-02-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain | interventions — Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All parties are masked other than the individual that will be dispensing the drug and preparing the medication (Placebo vs. Opioid).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid Group (Experimental): The participant will be plugged into an individualized comprehensive tiered pain plan that can include: Tier one (Acetaminophen, NSAIDS, Topicals, TENS unit, Massage, Acupuncture, Physical therapy. Tier two (Cognitive behavioral therapy, joint injections, nerve ablations, peripheral nerve stimulators) and less commonly Tier three (duloxetine, gabapentin). This is modeled after clinical practice. The participants will additionally receive prescription opioids for 6 weeks.
  Interventions: Drug: Opioid
- Placebo Group (Placebo Comparator): The participant will be plugged into an individualized comprehensive tiered pain plan that can include: Tier one (Acetaminophen, NSAIDS, Topicals, TENS unit, Massage, Acupuncture, Physical therapy. Tier two (Cognitive behavioral therapy, joint injections, nerve ablations, peripheral nerve stimulators) and less commonly Tier three (duloxetine, gabapentin). This is modeled after clinical practice. The participants will additionally receive a prescription opioid placebo for 6 weeks.
  Interventions: Drug: Opioid Placebo

INTERVENTIONS:
Drug: Opioid — Subjects will receive oral oxycodone as needed for pain which will be titrated weekly based on pain response, adverse effects, and patient preference. Subjects with intolerance to oxycodone will receive the equivalent dosing of morphine as an alternative.
  Arms: Opioid Group
Drug: Opioid Placebo — Subjects will receive a placebo capsule identical to oxycodone, which will similarly be titrated weekly. Subjects with intolerance to the first placebo will receive another placebo capsule identical to morphine.
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to determine whether exposure to prescription opioids is associated with brain structural changes on magnetic resonance imaging (MRI), with the primary outcome of white matter integrity as measured by fractional anisotropy of the corpus callosum.

DETAILED DESCRIPTION:
The investigators will recruit 200 adults aged 65 years and older with chronic pain of the knee or shoulder. Each will receive an individualized multimodal pain treatment pathway for 6-weeks - for half of participants this will include a prescription opioid; the other half will receive an identical placebo. After 6 weeks, participants will undergo opioid/placebo taper. The investigators will obtain neuroimaging (MRI), psychometric/cognitive testing, pain scores, and several exploratory patient-reported outcomes at several time-points: before the intervention (all tests), at 6 weeks (all tests except MRI), 6-month phone call (only phone based patient reported outcomes- no MRI), and at 1 year (all tests).

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* Pain for longer than 3 months (chronic)
* Moderate to severe pain nearly every day (averaged PEG score >5)
* Persistent pain despite use of >1 analgesic (Tylenol, Ibuprofen, lidocaine patch, etc)

Exclusion Criteria:

* Untreated severe/uncontrolled Mental health (schizophrenia, bipolar disorder, psychosis, history of suicidality, depression or anxiety, PTSD)
* Severe liver (cirrhosis) or kidney disease (ESRD on dialysis or GFR< 30)
* Cognitive impairment (Kokmen Short Test of Mental Status score < 29)
* Life expectancy < 12 months
* Contraindications to MRI
* Non-English speaking
* Opioid use within the past 6 months
* Contraindications or previous intolerance to prescription opioids
* Substance use disorder or high-risk for opioid-related adverse effects (Opioid Risk Tool ≥ 8)
* Residence outside of Minnesota or Wisconsin during opioid intervention period
* Another pain generator that is greater than their knee or shoulder or low back pain
* Anticipated surgery for joint replacement (Knee or shoulder) sooner than 3 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
White matter fractional anisotropy (FA) of corpus callosum | Baseline, 12 months
  Fractional anisotropy of the corpus callosum, adjusted against baseline value.

SECONDARY OUTCOMES:
White matter fractional anisotropy (FA) of other axonal tracts | Baseline, 12 months
  Fractional anisotropy of other white matter structures, adjusted against baseline value.
Gray matter cortical thickness | Baseline, 12 months
  Gray matter cortical thickness from major cortical regions, adjusted baseline values
Subcortical gray matter volumes | Baseline, 12 months
  Subcortical gray matter volumes on MRI, adjusted against baseline values
Mayo Preclinical Alzheimer's disease Cognitive Composite (Mayo-PACC) Global-z | Baseline, 6 weeks, 12 months
  This battery of tests includes AVLT (auditory verbal learning test), Animal Fluency, TMTB (trail making test B). Results are reported as a standardized z-score, where a higher z-score indicates better cognitive performance, with the score calculated by summing the z-scores of individual cognitive test components that make up the Mayo-PACC
Trailmaking Test A | Baseline, 6 weeks, 12 months
  Part A of the Trail Making Test consists of 25 numbered circles distributed over a sheet of paper. The participant is instructed to connect the circles in an ascending order, as quickly as possible, without lifting the pen or pencil from the paper. Results are reported as the number of seconds required to complete the task, higher scores indicate greater impairment.
Digit span memory test | Baseline, 6 weeks, 12 months
  The Digit Span memory test requires subjects to repeat series of digits of increasing length. Results are reported as the length of the longest correctly repeated sequence.
Mayo Test Drive | Baseline, 6 weeks, 6 month web based, 1 year
  Web based self-administered digital cognitive assessment focused on verbal memory, visual matching, and processing speed/executive function

CONTACTS AND LOCATIONS:
Overall Officials: Nafisseh Warner, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified summary measures will be made openly available to facilitate future scientific research from this NIA-supported effort. Deidentified individual level data will be available through a controlled access plan, which will require a confidential agreement and institutional review board (IRB) approvals as described in Element 5. MRI data will be linked to the cognitive measures as well as demographic information and clinical measures. In addition to numeric MRI outputs, raw or preprocessed MRI data will be made available in accordance with Brain Imaging Data Structure (BIDS) standards. Non-imaging data including psychometric testing and patient questionnaires will be available in raw form.
Supporting Information: Analytic Code
Time Frame: Scientific data will be deposited into the repository at the time of publication or the end of the award period, which comes first. Data will be preserved for a minimum of 5 years following the end of the grant period.
Access Criteria: De-identified datasets from this research study will be made available in accordance with the NIH Aging Research Biobank. Additional requests will be considered to the extent permissible under our IRB approvals, and local, state and federal laws and regulations, including the Privacy Rule. Additional requests for data should be directed to the study's Principal Investigators, who will evaluate the requests in a timely manner. Incoming proposals will be screened to ensure that the requests did not overlap or conflict with the funded efforts of this project. Approved requests will require a signed data use agreement and IRB approval to ensure that the usual procedures for participant protection are followed.